CLINICAL TRIAL: NCT01015066
Title: A Randomized Controlled Trial Comparing Buprenorphine/Naloxone With Naltrexone for Treatment in Opioid Dependent Adolescents and Young Adults
Brief Title: Comparison of Buprenorphine/Naloxone With Naltrexone in Opioid Dependent Adolescents
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study personnel left institution, anticipated funding did not occur
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Richard Blondell, MD, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMD04405009B
Record Dates: First submitted 2009-10-15; First posted 2009-11-17 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Opiate Addiction
Keywords: drug dependence; substance abuse; substance use disorders; buprenorphine; naltrexone; adolescents
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- buprenophine/naloxone (Active Comparator): Participants with this arm will receive 4-16 mg/d buprenorphine/naloxone (Suboxone).
  Interventions: Drug: Buprenorphine/naloxone
- Naltrexone (Experimental): Participants assigned to this arm will receive 50 mg/d naltrexone.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Sublingual tablets, 2/0.5mg (ratio buprenorphine:naloxone = 4:1), three times a day for six months (doses may be adjusted based on an individual's response)
  Other Names: Suboxone
  Arms: buprenophine/naloxone
Drug: Naltrexone — Oral tables, 50 mg/d, once a day for six months
  Other Names: ReVia
  Arms: Naltrexone

SUMMARY:
This study is designed to determine the relative effectiveness of buprenorphine/naloxone (Suboxone) pharmacotherapy versus naltrexone pharmacotherapy for treatment retention, relapse prevention and opioid craving reduction among opioid-dependent adolescents and young adults. The investigators hypothesize that naltrexone treatment is as effective as buprenorphine/naloxone for these treatment outcomes.

DETAILED DESCRIPTION:
Context: Standard treatment of opioid dependence in adolescents is detoxification and counseling, which results in relapse in 20-50% of patients. Alternative medical treatments include buprenorphine and naltrexone that have not been well investigated in adolescents and young adults. Buprenorphine has previously been shown effective in the treatment of opioid dependence in adolescents in one study in the United States as compared to detoxification. Although naltrexone treatment results in low compliance in adults, it is effective in combination with a strong social support network that exists in adolescents that live with at least 1 parent/guardian.

Objective: To compare the efficacy of buprenorphine/naloxone pharmacotherapy with naltrexone pharmacotherapy on treatment retention, relapse prevention and craving reduction among opioid-addicted adolescents and young adults.

Design: 2-arm Randomized Comparative Effectiveness Pharmacotherapy Clinical Trial.

Setting: The study will be conducted in an outpatient treatment facility Participants: The participants will be those who 1) are between 16-25 years old, 2) have clear evidence of a substance use disorder with opioid dependence, and 3) live with at least one parent.

Baseline data collection: Data collected at baseline will include (with examples), demographics (age, gender, race), substance use history (type of substances used, duration of use, routes of abuse), co-existing medical problems (seizures, hepatitis C), prior mental health problems (prior treatment, diagnoses), prior substance abuse treatment (outpatient, inpatient), socioeconomic variables (educational level, occupation, employment history), criminal history (number of arrests and convictions, total amount of time spent in jail or prison), family history (first degree relatives with substance use disorders) and scores on psychometric testing (DAST, opioid craving score).

Outcome data: Four main outcomes will be examined: Retention in treatment, self-reported opioid craving, self-reported drug use with urine toxicology confirmation. Retention in treatment (1-180 days) will be measured by the date that participant was last seen by study personnel or date when participant completes study following the date of enrollment. Opioid carving (1-10) will be measured by a 10 point visual analog scale. Self-reported drug use (days to first use and percent days abstinent) will be measured by time line follow back. Urine toxicology (yes/no) will be determined at baseline and monthly at 1, 2, 3, 4, 5, 6 months follow-up.

Data analysis: Outcome variables will be compared between the two groups using t-tests or chi-square tests as appropriate. A Kaplan-Myer survival analysis will be used to describe participant participation. Predictors of poor outcomes will be identified using a case-control design in which those with poor outcomes (the "cases") will be compared to those with successful outcomes (the "controls") using multivariate techniques (logistic regression).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Opiate Dependence
* Successful completion of detoxification
* can answer 9 out of 10 question correctly that tests understanding of the study

Exclusion Criteria:

* unable to pay for medication
* not living with a parent/guardian
* inability of patient and/or parent to give consent
* major co-occurring psychiatric disorder
* existing medical condition that would interfere with the treatment
* use of CNS depressants
* pregnancy

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Retention in treatment: (1-180 days) as measured by the date that participant was last seen by study personnel or date when participant completes study following the date of enrollment. | 6 months

SECONDARY OUTCOMES:
Opioid craving: (1-10) as measured by a 10 point visual analog scale. | 6 months
Self-reported drug use: (days to first use and percent days abstinent) as measured by time line follow back. | 6 months
Urine toxicology: (yes/no) at baseline and monthly at 1, 2, 3, 4, 5, 6 months follow-up. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Blondell, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- UB Department of Family Medicine, Buffalo, New York, United States